CLINICAL TRIAL: NCT01078012
Title: Pilot Study of Short Intervention for Medication Overuse Headache in General Practice
Brief Title: Short Intervention for Medication Overuse Headache (MOH) - Pilot
Acronym: SIMOHpilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Collaborators: Department of General Practice and Community Medicine, Oslo (Unknown); Head and Neck Research Group, Lørenskog (Unknown)
Responsible Party: Principal Investigator, Christofer Lundqvist, Principal Investigator, University Hospital, Akershus
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: SIMOH pilot
Record Dates: First submitted 2010-03-01; First posted 2010-03-02 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Medication Overuse Headache
MeSH Terms: conditions — Headache Disorders, Secondary

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Trained counselling (Active Comparator): Comparison of outcomes before intervention vs. 2 months after
  Interventions: Behavioral: Trained counselling

INTERVENTIONS:
Behavioral: Trained counselling

SUMMARY:
The purpose of the study is together with the BIMOH (NCT01314768) RCT study to evaluate whether training of GPs in the detection and treatment of medication overuse headache leads to improved care for these patients as compared to "business as usual".

DETAILED DESCRIPTION:
The present pilot study focuses on testing the logistics and the methodology of short intervention on a pilot group of GPs and their patients.

Due to low recruitment and the pilot study focus on logistics and methodology, the study was changed to not include a control (business as usual) arm. The outcomes were evaluated as "before - after" data and qualitative comments on acceptability and utility of the method. Primary outcomes were changed to be the acceptability and utility (previously listed as secondary outcomes) while secondary outcomes were headache days and medication days (previously listed as primary).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with medication overuse headache

Exclusion Criteria:

* Other complicating pain condition

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2010-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Qualitative comments of participants on acceptability and utility | 2 months

SECONDARY OUTCOMES:
Qualitative comments of participants on acceptability and utility. | 2 months
Number of medication days per month | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General Practice and Community Medicine, Oslo, Oslo County, Norway

REFERENCES:
- [Derived] Kristoffersen ES, Straand J, Russell MB, Lundqvist C. Feasibility of a brief intervention for medication-overuse headache in primary care--a pilot study. BMC Res Notes. 2014 Mar 20;7:165. doi: 10.1186/1756-0500-7-165. PMID 24646429